CLINICAL TRIAL: NCT06675344
Title: A Randomized, Double-blind, Clinical Trial of the Apollo Device in Systemic Sclerosis for the Management of fatiguE, Raynaud Phenomenon and qualiTy of Life (ASScERT-QoL)
Brief Title: The Apollo Device in Systemic Sclerosis for the Management of fatiguE, Raynaud Phenomenon and qualiTy of Life
Acronym: ASScERT-QoL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Robyn T. Domsic, MD, MPH (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Robyn T. Domsic, MD, MPH, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY24040026; HT94252410456 (Other Grant/Funding Number: U.S. Department of Defense)
Record Dates: First submitted 2024-10-30; First posted 2024-11-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Systemic Sclerosis (SSc)
Keywords: Scleroderma; Raynaud Phenomenon; fatigue
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Raynaud Disease; Fatigue

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, sham device-controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Apollo Neuro Device (Experimental): Apollo Neuro Device
  Interventions: Device: Apollo Neuro Device
- Sham Device (Sham Comparator): Study participants will be randomized 1:1 (Apollo Neuro device : Sham device) Devices are identical; however, the sham device will be set to a frequency that has no therapeutic benefits.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Apollo Neuro Device — The Apollo Neuro wearable device is an Apple Watch-sized wearable device that delivers vibration at set frequencies , termed transcutaneous vibratory stimulation, or TVS. These low volume sound waves feel like a soothing touch to the skin (TVS) and activate touch receptors. Apollo is controlled via smartphone and worn on the wrist or ankle. The Apollo is fitted with an adjustable band, made of a durable neoprene material with polyester overlays. Participants are asked to wear it daily for a minimum time period for 6 weeks. Users can choose from different modes of vibration, with some being energizing, others relaxing.
  Arms: Apollo Neuro Device
Device: Sham device — The Apollo Neuro is an Apple Watch-sized wearable device that delivers vibration, termed transcutaneous vibratory stimulation, or TVS. The sham device is identical in appearance to the active intervention, but provides a lower frequency vibration that has no known therapeutic benefit.
  Arms: Sham Device

SUMMARY:
The purpose of this study it to test the efficacy of a wearable device to improve symptom management and maximize qualify of life in systemic Sclerosis (SSc) patients in a randomized trial. Specifically, we will evaluate if the Apollo Neuro device may improve the two specific symptoms highest ranked by patients as affecting qualify of life (fatigue, Raynaud phenomenon) as co-primary outcomes.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a multisystem autoimmune disease that is characterized by progressive vasculopathy, excessive fibrosis, and immune system activation. Fatigue in SSc is common and greatly impacts quality of life: The prevalence of fatigue in SSc patients is significantly higher than the general population. Raynaud phenomenon (RP) in SSc is not only the most common SSc manifestation, affecting nearly all but is often the earliest SSc symptom. SSc-RP is the highest ranked SSc-related symptom affecting quality of life, and is a major cause of SSc-related morbidity. There are currently no approved medications to treat RP, SSc-associated RP phenomenon or fatigue in SSc. Thus, a non-pharmacologic intervention has the potential to provide SSc patients with a new treatment modality without common limiting side effects, and access. The Apollo wearable provides transcutaneous vibratory stimulation, and can be worn on the wrist or ankle.

Goal: To recruit 160 SSc patient participants into this randomized, sham-device controlled clinical trial. Patients will be randomized 1:1 to receive the Apollo vs. sham wearable, which they will wear daily for 6 weeks.

Outcome measures focus on quality-of-life.

.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Ability to provide written informed consent,
3. Diagnosis of SSc, as defined by the 2013 ACR/EULAR classification of SSc64 with a positive ANA
4. Baseline score ≥55 on the FACIT-Fatigue scale,
5. Presence of Raynaud phenomenon with ASRAP-SF severity of T-score ≥40,
6. Steady daily doses and any immunosuppressive medication, vasodilators or other medications used to treat pulmonary hypertension, antidepressants and anxiolytic use for 4 weeks prior to baseline
7. Currently owns and operates an iOS or Android smart phone regularly
8. Ability to comply with the clinical visits schedule and the study-related procedures.

Exclusion Criteria:

1. History of sympathectomy or stellate ganglion block
2. History of Botox injections to the digits within the last 3 months
3. Diabetes mellitus
4. Major surgery within 8 weeks
5. Hospitalization for any reason within four weeks of the study baseline visit
6. Active malignancy
7. Pregnant or breastfeeding women,
8. End-stage renal disease (estimated glomerular filtration rate < 15 mL/min/1.73m2) or on dialysis,
9. Hepatic insufficiency as defined by function worse than Child-Pugh Class B
10. Medication exclusions:

    1. actively prescribed standing doses of beta-blockers,
    2. actively prescribed standing doses of sedatives, hypnotics, opioids, benzodiazepines or anti-psychotic medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue | Baseline, 6 Weeks
  The PROMIS® (Patient-Reported Outcomes Measurement Information System) SF v1.0 Fatigue 13a scale. This is a13-item, patient reported measure of an individual's level of fatigue during their usual daily activities over the past week. The raw score is converted to a T-score for analysis with 50 for the mean and a standard deviation of 10.
Change in average weekly Raynaud attacks | Baseline, 6 Weeks
  Average number of weekly Raynaud attacks. Over a period of one week, patients will record their Raynaud phenomenon (RP) attack frequency via a smartphone app. The Raynaud app is usable on both Apple iPhones and Android phones.

SECONDARY OUTCOMES:
Change in quality of life | baseline up to week 6
  The EuroQol (EQ)-5D-5L will be used. The quality-of-life assessment instrument has 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a patient global assessment visual analog scale (VAS). In the EQ-5D-5L each dimension is ranked on 5 levels of severity. Full health is a score of 1 and values below zero are regarded as a state worse than death.
Change in Raynaud phenomenon symptom severity | baseline to week 6
  The ASRAP (Assessment of Scleroderma-associated RAynaud's Phenomenon) Questionnaire Short form is a 10-item patient self-report questionnaire regarding symptoms over the last week. Raw scores are converted to T-score with a median of 50.
Change in the Raynaud Condition Score | baseline to week 6
  The Raynaud Condition Score is a patient-reported outcome of a single question regarding Raynaud severity. It is a visual analog scale with a results range of 0-100. A score of 0 is no symptoms, and 100 is severe symptoms. It is recommended by OMERACT for assessment of Raynaud phenomenon.
Change Sleep | change from baseline to week 6
  PROMIS® Sleep disturbance short form 4a will be used. This 4-item questionnaire uses a 5-point Likert scale for responses, inquiring about symptoms over the last week. Raw scores are converted to T-scores, with a mean of 50 and SD of 10.
Change in pain | baseline to week 6
  We will use the PROMIS pain interference (v1.1- Short Form 4a) questionnaire which poses 4 questions regarding the last week of pain symptoms. Responses are in a 5-point likert scale from not at all to very much. Raw scores are converted to T-scores for analysis with a median of 50 and standard deviation of 10.
Change in depression | change baseline to week 6
  Depression as measured by the Patient Health Questionnaire (PHQ-8). These 8 questions are responded to with a Likert scale of 0(never) up to 3 (always) with a score range of 0-27.
Change in Social Function | baseline to week 6
  Captured using PROMIS Short Form v2.0 - Ability to Participate in Social Roles and Activities 4a. This is a 4-question survey, with respondents answering a 5-point likert scale from 'never' to 'always'. Raw scores are converted to T-scores with a mean of 50 and standard deviation of 10.
Change in dysautonomia symptoms | baseline to week 6
  Change in dysautonomia symptoms as measured with the COMPASS-31 scale. This is a 31-question instrument which includes six domains: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder and pupillomotor . A higher score indicates worse autonomic function. Following appropriate weighting, this instrument provides an autonomic symptom score from 0 to 100.
Change in pain intensity | baseline to week 6
  PROMIS® Numeric Rating Scale v.1.0 - Pain Intensity 1a will be used. This is a single question inquiring about pain in the last week, rating from 0 (no pain) to 10 (worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Robyn T Domsic, MD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - DelRicht Research Center, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - University of Pittsburgh and UPMC Scleroderma Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Requests for IPD can be obtained by emailing the PI of the study.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available after the study has been completed and published
Access Criteria: We will comply with the CDMRP policy for data sharing, while also complying with all pertinent local, state, and federal regulations. All individuals requesting the data sets will be required to enter into a data share agreement that: (1) acknowledges that the data will be stripped of any identifying markers, (2) acknowledge the data will only be utilized for research purposes, and (3) assure that the requesting investigator will destroy the raw data when the research is completed.

REFERENCES:
- [Background] Yu L, Domsic RT, Saketkoo LA, Withey J, Frech TM, Herrick AL, Hummers LK, Shah AA, Denton CP, Khanna D, Pauling JD. Assessment of the Systemic Sclerosis-Associated Raynaud's Phenomenon Questionnaire: Item Bank and Short-Form Development. Arthritis Care Res (Hoboken). 2023 Aug;75(8):1725-1734. doi: 10.1002/acr.25038. Epub 2023 Jan 30. PMID 36214062